CLINICAL TRIAL: NCT01790711
Title: The Efficiency of Fecal Microbiota Transplantation on Type 2 Diabetes Mellitus
Brief Title: Fecal Microbiota Transplantation on Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Vice chief, medical center for digestive diseases, The Second Hospital of Nanjing Medical University
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMT-CN-121025
Record Dates: First submitted 2013-02-09; First posted 2013-02-13 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Efficiency; Methodology
Keywords: Gut bacteria; Bacteria; Fecal transplant; Bacteriotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FMT by endoscopy (Experimental): Once, fresh or frozen bacteria
  Interventions: Procedure: FMT through mid-gut

INTERVENTIONS:
Procedure: FMT through mid-gut
  Other Names: FMT through mid-gut by gastroscope

SUMMARY:
The gut microbiota is considered to constitute a "microbial organ" which has pivotal roles in the body's metabolism. Evidence from animal and human studies strongly support the link between intestinal bacteria and type 2 diabetes mellitus. The present clinical trial aims to re-establish a gut functionality state of intestinal flora through fecal microbiota transplantation.

DETAILED DESCRIPTION:
We established a standard bacteria isolation from donated fresh stool in lab.Then the bacteria is transplanted to mid-gut (at least below the second part of duodenum ) through regular gastroscope. Participants in this study will be randomly assigned to receive fecal microbiota transplantation only once or traditional therapy, and accept follow-up for at least one year. Blood tests,OGTT and magnetic resonance spectroscopy will be used to assess participants at study start and at study completion.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes mellitus

Exclusion Criteria:

With any cause of liver disease other than fatty liver Known or suspected cirrhosis Inability or unwillingness to undergo OGTT and magnetic resonance procedures Requirement of long-term antibiotic therapy Pregnancy, breast-feeding, or plans to become pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-05 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
The Efficiency of FMT on T2DM | Up to 24 months
  Confirmed by the tests of blood glucose level, OGTT, HACb1 and C-peptide.

SECONDARY OUTCOMES:
Durability | Up to 12 months
  Measure the durability of the therapy effects.Based on the tests of blood glucose level, HACb1 and C-peptide. BMI also will be observed.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Vrieze A, Van Nood E, Holleman F, Salojarvi J, Kootte RS, Bartelsman JF, Dallinga-Thie GM, Ackermans MT, Serlie MJ, Oozeer R, Derrien M, Druesne A, Van Hylckama Vlieg JE, Bloks VW, Groen AK, Heilig HG, Zoetendal EG, Stroes ES, de Vos WM, Hoekstra JB, Nieuwdorp M. Transfer of intestinal microbiota from lean donors increases insulin sensitivity in individuals with metabolic syndrome. Gastroenterology. 2012 Oct;143(4):913-6.e7. doi: 10.1053/j.gastro.2012.06.031. Epub 2012 Jun 20. PMID 22728514
- [Background] Koren O, Goodrich JK, Cullender TC, Spor A, Laitinen K, Backhed HK, Gonzalez A, Werner JJ, Angenent LT, Knight R, Backhed F, Isolauri E, Salminen S, Ley RE. Host remodeling of the gut microbiome and metabolic changes during pregnancy. Cell. 2012 Aug 3;150(3):470-80. doi: 10.1016/j.cell.2012.07.008. PMID 22863002
- [Background] Borody TJ, Khoruts A. Fecal microbiota transplantation and emerging applications. Nat Rev Gastroenterol Hepatol. 2011 Dec 20;9(2):88-96. doi: 10.1038/nrgastro.2011.244. PMID 22183182
- [Background] Aroniadis OC, Brandt LJ. Fecal microbiota transplantation: past, present and future. Curr Opin Gastroenterol. 2013 Jan;29(1):79-84. doi: 10.1097/MOG.0b013e32835a4b3e. PMID 23041678
- [Background] Zhang F, Luo W, Shi Y, Fan Z, Ji G. Should we standardize the 1,700-year-old fecal microbiota transplantation? Am J Gastroenterol. 2012 Nov;107(11):1755; author reply p.1755-6. doi: 10.1038/ajg.2012.251. No abstract available. PMID 23160295
- See also: Fecal microbiota transplantation — http://www.ncbi.nlm.nih.gov/pubmed